CLINICAL TRIAL: NCT03604653
Title: Trial of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Primary Peritoneal Cancers and Secondary Peritoneal Cancers From Stomach, Colorectal, Appendiceal, and/or Gynecological Origins
Brief Title: Trial of Cytoreductive Surgery and HIPEC in Patients With Primary and Secondary Peritoneal Cancers
Status: Completed | Type: Observational
Sponsor: Holy Name Medical Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: holynameHIPEC1
Record Dates: First submitted 2018-07-12; First posted 2018-07-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Stomach Cancer; Colorectal Cancer; Appendiceal Cancer; Ovarian Cancer; Uterine Cancer; Cervical Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: HIPEC; Stomach cancer; colorectal cancer; appendiceal cancer; ovarian cancer; uterine cancer; cervical cancer; fallopian tube cancer; primary peritoneal carcinoma; intraperitoneal chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Appendiceal Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Mitomycin; Cisplatin; Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stomach: Heated Intraperitoneal Chemotherapy with Mitomycin C 30mg at time 0, 10mg at time 45 minutes, CDDP Cisplatin 50mg/m2@ time 0
  Interventions: Device: HIPEC; Drug: Mitomycin c; Drug: CDDP 50
- Colorectal, Appendiceal, Pseudomyxoma Peritonei: Heated Intraperitoneal Chemotherapy with Mitomycin C 30mg at time 0, 10mg at time 45 minutes
  Interventions: Device: HIPEC; Drug: Mitomycin c
- Primary Peritoneal: Heated Intraperitoneal Chemotherapy with CDDP Cisplatin 50mg/m2 at time 0, Doxorubicin 15mg/m2 at time 0
  Interventions: Device: HIPEC; Drug: CDDP 50; Drug: Doxorubicin
- Ovarian, Cervical, Uterine, Fallopian Tube: Heated Intraperitoneal Chemotherapy with CDDP Cisplatin 75mg/m2 at time 0
  Interventions: Device: HIPEC; Drug: CDDP 75

INTERVENTIONS:
Device: HIPEC — Heated chemotherapy is pumped into the abdomen and circulated for 90 minutes
  Other Names: Chemo bath
Drug: Mitomycin c — MMC 30mg@ T0, 10mg@T45 min
  Other Names: MMC
  Groups: Colorectal, Appendiceal, Pseudomyxoma Peritonei; Stomach
Drug: CDDP 50 — 50mg/m2@T0
  Other Names: Cisplatin
  Groups: Primary Peritoneal; Stomach
Drug: CDDP 75 — 75mg/m2@T0
  Other Names: Cisplatin
  Groups: Ovarian, Cervical, Uterine, Fallopian Tube
Drug: Doxorubicin — 15mg/m2@T0
  Other Names: DXR
  Groups: Primary Peritoneal

SUMMARY:
Patients with primary peritoneal cancer or secondary peritoneal cancers from stomach, colorectal, appendiceal, and gynecological primary origin will be screened by pathology and staging to see if they are eligible to undergo cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (HIPEC).

To be eligible for the study, patients must be over 18 years of age, have appropriate pathology and stage with disease confined to the peritoneal cavity, have a good performance status, have laboratory values that fall within safe ranges to undergo an operation and receive intraperitoneal chemotherapy. The chemotherapeutic agent and dose will be assigned based on pathological diagnosis in accordance with current standard of care.

Surgery will be performed with the goal of removing all visible tumor that may require removal of adjacent organs. Once only microscopic disease is present, the chemotherapy will be delivered directly into the peritoneum via intraperitoneal hyperthermia and perfusion device. This will continue for 90 minutes.

Patients will be followed for tumor response, survival, toxicity, complications, quality of life, and tumor markers. They will have regular follow up visits with the surgeon, undergo routine surveillance imagings, and receive follow up phone calls periodically.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis can be caused by primary peritoneal cancers and secondary peritoneal spread from stomach, colorectal, appendiceal, and/or gynecological cancers. Combined presentation of patients with peritoneal carcinomatosis make up about 67,000 new cancer diagnoses each year. Of these cases, about 25,000 patients are estimated to be candidates for cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (HIPEC); however, in 2009 only five percent of these patients received such treatment.

Alternative therapies to cytoreductive surgery and HIPEC are few. They include surgical treatments with cytoreduction alone which are palliative in nature and inadequate to manage the disease, radiation which is limited in regard to tumors disseminated throughout abdominal cavity, systemic chemotherapy which has poor penetration into the peritoneum. Intraperitoneal chemotherapy via indwelling peritoneal catheter is limited due to port infections, toxicity, and unequal distribution in the abdominal cavity.

For patients whose disease is limited to the peritoneal cavity, multi-modality treatment with cytoreductive surgery followed by intraoperative HIPEC can deliver chemotherapy directly to microscopic tumors at a higher concentration than is tolerated systemically. It causes disruption of cell membranes and induces apoptosis. Moreover when intraperitoneal chemotherapy is given at a higher temperature, it has a selective lethal effect on cancer cells secondary to improved tissue absorption. The typical side effects of systemic chemotherapy are also minimized with HIPEC.

HIPEC is given intraoperatively in one treatment setting after all visible disease has been resected (i.e., cytoreductive surgery). The goal of cytoreductive surgery is to leave behind only microscopic disease and may require removal of adjacent organs. HIPEC is then delivered via tubings with temperature probes that are placed in the intraperitoneal cavity. The skin is then temporarily closed and the tubings are connected to a intraperitoneal hyperthermia and perfusion device that delivers sterile solution with chemotherapy into the abdomen. The device heats and circulates the chemotherapy for 90 minutes. After HIPEC is completed, abdomen is reopened and copiously irrigated. Surgical reconstruction with any removed organs (such as bowel) and fascial/skin closure are the final steps.

Previous studies have shown conflicting results on survival benefit for patients with some of the aforementioned secondary peritoneal cancers who have undergone cytoreductive surgery and HIPEC. This study is an outcomes based study that seeks to look at the impact of HIPEC on overall survival and recurrence-free survival.

ELIGIBILITY:
Inclusion Criteria:

Age >18

Diagnosis at the time of resection or on frozen section of:

* recurrent or primary stomach, colorectal or appendiceal cancer with regional spread that is confined to the peritoneal cavity
* primary peritoneal cancer
* ovarian cancer stage IC or higher
* uterine or cervical cancer stage IIA or higher with recurrence confined to the peritoneum
* fallopian tube cancer stage III or recurrence confined to the peritoneum ECOG performance status of 0,1, or 2

Lab values:

* absolute neutrophil count >1500
* platelets >100,000
* creatinine less than or equal to 2.0mg/dL
* bilirubin less than or equal to 1.5 times the upper limit of normal
* SGOT and alkaline phosphatase less than or equal to 2.5 times the upper limit of normal
* patients of childbearing age must have a negative serum pregnancy test and be using an effective form of contraception

Exclusion Criteria:

* Extra-peritoneal disease or unresectable disease
* Any known sensitivity to the chemotherapeutic agents used in the study
* Significant medical comorbidities that would prevent the patient from being able to complete the protocol (at discretion of investigator)
* Patients with gynecological malignancy who desire future fertility
* An informed consent cannot be obtained from the patient or power of attorney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary peritoneal cancers and secondary peritoneal cancers from stomach, colorectal, appendiceal, and/or gynecological origins who are eligible by stage and pathology for surgical debulking and HIPEC, and who meet criteria to undergo an extensive operation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to 10 years
  Time from HIPEC treatment to death
Disease-free Survival | up to 10 years
  Time from HIPEC treatment to either recurrence or relapse of cancer, or death

SECONDARY OUTCOMES:
Complications | 90 Days
  Patients who undergo cytoreductive surgery followed by HIPEC will be monitored to record the incidence of the following complications: fistula, leak, pulmonary embolus, deep vein thrombosis, re-operation, hematologic
Treatment related quality of life changes as measured by the WHO QOL-BREF questionnaire | Up to 10 years
  Treatment related quality of life changes will be measured by the WHO QOL-BREF at each follow up visit
Tumor Markers | up to 10 years
  Cancer-specific tumor markers will be measured 6 months post operatively and then yearly.
Toxicity as measured by treatment related adverse events according to the NCI CTCAE v 4.0 | 90 Days
  Toxicity as measured by adverse events grade III-V according to NCI CTCAE v.4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No